CLINICAL TRIAL: NCT00225901
Title: Phase I/II Study of Recombinant Human Hepatocyte Growth Factor in Fulminant and Late-Onset Hepatic Failure
Brief Title: Phase I/II Study of Recombinant Human Hepatocyte Growth Factor in Fulminant Hepatic Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRC02HG-I/II-1
Record Dates: First submitted 2005-09-21; First posted 2005-09-26 (Estimated); Last update posted 2005-09-26 (Estimated); Status verified 2005-09

CONDITIONS: Liver Failure, Acute
MeSH Terms: conditions — Liver Failure, Acute

INTERVENTIONS:
Drug: Recombinant human hepatocyte growth factor

SUMMARY:
The purpose of this study is to determine whether recombinant human hepatocyte growth factor is safe and effective in the treatment of fulminant and late-onset hepatic failure.

DETAILED DESCRIPTION:
Fulminant and late-onset hepatic failure (LOHF) is intractable disease with high degree of fatality (70-80%). Only liver transplantation is established as a therapeutic modality to rescue patients with fulminant hepatic failure or LOHF. However, approximately 75% of the patients are not able to receive liver transplantation in Japan, and effective non-surgical treatment has not been established yet. Hepatocyte growth factor (HGF) is one of major agents stimulating liver regeneration and ameliorating hepatic injury.

In this study, recombinant human HGF is administered to patients with fulminant hepatic failure or LOHF, who can not receive liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fulminant or late-onset hepatic failure
* Must be unable to receive liver transplantation

Exclusion Criteria:

* Under 16 years old
* Cancer patients
* Pregnancy-aged women
* Impaired renal function
* Impaired cardiac function
* Severe complications including pneumonia, sepsis, DIC and so on

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2005-09

PRIMARY OUTCOMES:
All adverse effects throughout the protocol

SECONDARY OUTCOMES:
Survival time at 4 weeks
Degree of hepatic encephalopathy at 3, 5, 8, 11, 15, 21, and 28 days
Liver function test at at 3, 5, 8, 11, 15, 21, and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Chiba, M.D., Principal Investigator — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan